CLINICAL TRIAL: NCT06620367
Title: Innovative Approach in Guided Bone Regeneration Using Digitally Designed Surgical Guide
Brief Title: Guided Sausage Technique in Bone Regeneration As a Novel Digital Work Flow
Acronym: RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mona Al-Ahmady El-Meligy, lecturer of periodontology, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #R-OMPDR- 6-24-3122
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Digital Guided Bone Regeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional guided bone regeneration (Active Comparator): a medium horizontal ridge defect will receive bone graft and covered with membrane
  Interventions: Procedure: conventional guided bone regeneration
- digital guided bone regeneration (Active Comparator): digital designed guide will be used in a medium horizontal ridge defect to place bone graft and covered with membrane
  Interventions: Procedure: digital guided bone regeneration

INTERVENTIONS:
Procedure: conventional guided bone regeneration — 10 sites with medium horizontal ridge defect will be treated with bone graft (50%autogenous mixed with 50%xenograft) covered with bilayer collagen membrane stabilized by tacks
  Arms: conventional guided bone regeneration
Procedure: digital guided bone regeneration — 10 sites with medium horizontal ridge defect will be treated with bone graft (50%autogenous mixed with 50%xenograft) placed by digital designed guide covered with bilayer collagen membrane stabilized by tacks
  Arms: digital guided bone regeneration

SUMMARY:
The goal of this clinical trial is to compare amount of bone resorption and flap dehiscence following guided bone regeneration with or without digitally designed surgical guide. The main questions it aims to answer are:

* Does it differ in amount of bone resorption between the conventional and digital guided bone regeneration?
* What is the difference between conventional and digital protocols regarding flap dehiscence following guided bone regeneration? Researchers will compare digital guided versus conventional technique to choose adequately which protocol to use.

Participants will:

* Receive guided bone regeneration around implant
* Visit the clinic after 2,7,14 days for detection any signs of flap dehiscence
* Bone gain and bone density will be assessed after 6 months

DETAILED DESCRIPTION:
Twenty sites with ridge defects will be recruited for this study. All investigations will be carried out in accordance with the 1975 Helsinki Declaration, as revised in 2013 for clinical approval. The purpose of the present study will be explained to the patients and informed consents will be obtained . Sites were randomly divided into 2 treatment groups .10 sites will be treated with bone graft (50%autogenous mixed with 50%xenograft) covered with bilayer collagen membrane without use of guide & 10 sites will receive the same treatment except it will be guided using digitally designed guide. Membranes in both groups will be stabilized by tacks. Following clinical parameters will be recorded: the wound opening of buccolingual distance between sutured flap margins with a UNC periodontal probe to the nearest millimeter at 2, 7 and 14 days, flap dehiscence. Also, bone gain and bone density will be assessed using cone beam computed tomography (CBCT) at baseline and 6 months post-surgery. The collected data was statistically analyzed at the different follow up periods.

ELIGIBILITY:
Inclusion Criteria:

* medium horizontal ridge defect according to clone classification
* must have a general health showing no contraindications for surgery
* must be at least 35 years old
* patients also have adequate soft tissue thickness and width of keratinized gingiva

Exclusion Criteria:

* no sign of uncontrolled systemic diseases
* non smoker
* not pregnant
* sever ridge deficient
* patients below 18 years old

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-09-24 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
flap dehiscence | 14 days
  the flap dehiscence will be assessed using a UNC periodontal probe through the the wound opening of buccolingual distance between sutured flap margins

SECONDARY OUTCOMES:
bone gain | 6 months
  bone gain will be assessed using cone beam computed tomography (CBCT)
bone denisty | 6 months
  cone beam computed tomography (CBCT) will be used to asses bone density

CONTACTS AND LOCATIONS:
Overall Officials: Bassem nabil elfahl, assistant professor, Principal Investigator — faculty of dentistry Tanta university
Locations (1):
- faculty of dentistry Tanta university, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No